CLINICAL TRIAL: NCT05058313
Title: Evaluation of the Safety and Performance of the MILTA GYNECO Vaginal Probe in Postmenopausal Women With Vaginal Atrophy Resistant to All Non-invasive Therapies for More Than 3 Months - Pilot Study of First Use in Females
Brief Title: Evaluation of the Safety and Performance of the MILTA GYNECO Vaginal Probe in Postmenopausal Women With Vaginal Atrophy
Acronym: SIVAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: PHYSIOQUANTA (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDIL/2020/PM-001
Record Dates: First submitted 2021-08-27; First posted 2021-09-27 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Menopause; Urinary Incontinence; Atrophic Vaginitis
Keywords: post-menopausal period; low level light therapy; genitourinary
MeSH Terms: conditions — Urinary Incontinence; Atrophic Vaginitis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postmenopausal patients (Experimental)
  Interventions: Device: Photobiomodulation

INTERVENTIONS:
Device: Photobiomodulation — Six weekly photobiomodulation sessions (PBMT) using the MILTA ™ GYNECO vaginal probe.

SUMMARY:
Vulvovaginal atrophy is common after menopause, with a significant negative effect on quality of life. Large cohort studies have reported the prevalence of vaginal dryness to be between 27% and 55% and dyspareunia between 32% and 41%. Management of urogenital atrophy includes lifestyle modification, nonhormonal treatments (vaginal lubricants or moisturizers, laser treatments), as well as hormonal treatments. The disadvantages of the non-surgical methods are average results, discontinuation, and frequent contraindications to hormonal treatments.This has led to a strong interest in the development of non-invasive or minimally invasive methods that are easy to implement, effective and durable.

Photobiomodulation therapy (PBMT) has been proposed as an alternative for the treatment of genitourinary menopausal syndrome (GMS) and stress urinary incontinence. PBMT devices exert their effect via non-thermal mechanisms. PBMT stimulates collagen and elastin synthesis in the vaginal tissue, to support the urethrovaginal sphincter and urethra, and to promote vasodilation in the vaginal and urethral submucosa. PHYSIOQUANTA has developed a vaginal probe coupled with its innovative MILTA™ process synergistically combining NPCL (Nano-Pulsed Cold Laser) laser emitters, infrared diodes and RGB (Red Green Blue) diodes, operating in a magnetic tunnel. The MILTA acts deeper than LEDs, due to the diffusion of photons in soft tissues.

In this study, the study investigators aimed to evaluate the safety and performance of the MILTA™ GYNECO vaginal probe in a pilot study of first use in women. This clinical study on the MILTA vaginal probe is expected to result in its CE marking Class IIb DM.

ELIGIBILITY:
Inclusion Criteria:

* Patient with pelvic discomfort/pain (pain, dryness, irritation, etc.) due to vaginal atrophy that has failed all non-invasive therapies for over 3 months.
* Postmenopausal patient recruited during a consultation in the Gynecology department of the University Hospital of Nîmes or at the KARIS Medical Center in Perpignan and having undergone a complete clinical examination allowing any physical and / or psychological cause to be eliminated.
* Patient who has given her free and informed consent.
* Patient affiliated or beneficiary of a health insurance plan.

Exclusion Criteria:

* Patient not available for the 6-week follow-up.
* Patient presenting with pelvic pain of physical and / or psychological origin.

  * Patients undergoing initial treatment for cancer and/or who have completed their treatments within the last year
  * Patient with immunosuppression.
  * Allergy to the material of the probe protection used (latex for example).
* Pregnancy.
* Implantable device active in the heart such as a defibrillator or a pacemaker, neuromodulation stimulator, electrodes implanted for the treatment of Parkinson's disease.
* Epilepsy, photophobia, recent intake of photosensitizing drugs or cosmetics (in the last 6 months), history of porphyria.
* Patient participating in category 1 interventional study.
* Patient in an exclusion period determined by another study.
* Patient under legal protection, under guardianship or under curatorship.
* Patient for whom it is impossible to give informed information.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Day 1
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Week 1
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Week 2
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Week 3
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Week 4
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Week 5
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] of the use of the MILTA™ GYNECO vaginal probe | Week 6
  Collection and investigation of the causality of adverse events linked to the treatment (expected adverse effects: burns, pain on penetration, tingling, edema, allergic reaction).

SECONDARY OUTCOMES:
Performance of the MILTA™ GYNECO vaginal probe on pain linked to vaginal atrophy | Day 0
  Visual analogue scale (0-10): the device will be considered effective if the VAS pain score decreases by at least 30%
Performance of the MILTA™ GYNECO vaginal probe on pain linked to vaginal atrophy | Week 6
  Visual analogue scale (0-10): the device will be considered effective if the VAS pain score decreases by at least 30%
Performance of the MILTA™ GYNECO vaginal on the vaginal mucosa | Day 0
  Vaginal Health Index: Score 1-5
Performance of the MILTA™ GYNECO vaginal on the vaginal mucosa | Week 6
  Vaginal Health Index: Score 1-5
Vaginal pH | Day 0
  pH value between 4 - 7.5
Vaginal pH | Week 6
  pH value between 4 - 7.5
Vaginal flora | Day 0
  Nugent score: score from 0 to 10: 0 to 3: normal flora predominantly lactobacilli, 4 to 6: intermediate flora with scant lactobacilli and associated with other poorly differentiated bacterial morphotypes in small quantities, 7 to 10: suggestive of bacterial vaginosis
Vaginal flora | Week 6
  Nugent score: score from 0 to 10: 0 to 3: normal flora predominantly lactobacilli, 4 to 6: intermediate flora with scant lactobacilli and associated with other poorly differentiated bacterial morphotypes in small quantities, 7 to 10: suggestive of bacterial vaginosis
Patient satisfaction Patient satisfaction | Week 6
  Patient Global Impression of Change (PGI-C): Patients will be classified into 3 categories according to their score: deterioration (score of 1 to 3), stable (score of 4), improvement (score of 5 to 7)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Mares, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (3):
- France (3):
  - CHU Nîmes, Nîmes
  - Centre Médical KARIS, Perpignan
  - Centre Hospitalier de Valenciennes, Valenciennes

REFERENCES:
- [Result] Salerno J, Serrand C, Kabani S, Chevallier T, de Tayrac R, Mares P. Safety and performance of photobiomodulation delivered by vaginal probe in patients with genitourinary syndrome of menopause. Climacteric. 2025 Dec 17:1-7. doi: 10.1080/13697137.2025.2591279. Online ahead of print. PMID 41404945